CLINICAL TRIAL: NCT06245720
Title: Serum and Urine Metabolome Studies in Patients With Acute Kidney Injury After Cardiac Surgery
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: KY20240123-01
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-01

CONDITIONS: Cardiac Surgery Associated Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — The serum sample was obtained by collecting blood samples with a serum separation hose containing serum procoagulant, allowing it to coagulate after standing at room temperature for 60min, centrifuging at 3000rmb at 4 °C for 10 min, aspirating the supernatant (i.e., serum 200ul) and dividing it into a suitable numbered 2ml centrifuge tube, liquid nitrogen quick-freezing for 5-10 min, and storage in a -80 °C freezer to avoid repeated freezing and thawing. Urine specimen collection is to use urine in a urine bag, centrifuge at 10000rmb at 4 °C for 10min, aspirate 500ul of supernatant in a numbered 2ml sterile centrifuge tube, liquid nitrogen quick-freeze for 5-10min, and store in a freezer at -80 °C to avoid repeated freezing and thawing.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AKI group: AKI is then defined as an increase in serum creatinine (SCr) of at least 26.4 μmol/L over 48 hours, or an increase in SCr greater than 1.5 times baseline over 7 days, or a urine output of less than 0.5 mL/kg per hour for more than 6 hours, according to the Kidney Disease: Improving Global Outcomes (KDIGO) guidelines.
- Non-AKI group: According to the Kidney Disease: Improving Global Outcomes (KDIGO) guidelines, patients do not develop acute kidney injury.

INTERVENTIONS:
Other:

SUMMARY:
The goal of this observational study is to learn about serum and urine metabolome in patients after cardiac surgery.

DETAILED DESCRIPTION:
The main objective of this study is to collect blood and urine samples from patients after cardiac surgery, and to perform metabolomic analysis to find the differential metabolites and their enrichment pathways in AKI patients and non-AKI patients.The secondary objective is to intervene in its enrichment pathway to find ways to improve CSA-AKI.

ELIGIBILITY:
Inclusion Criteria:

1. Age> 18 years old;
2. after cardiopulmonary bypass;

Exclusion Criteria:

1. Under the age of 18;
2. Previous chronic kidney disease or receiving renal replacement therapy;
3. Have a history of kidney transplantation or nephrectomy.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with cardiac surgery who have undergone cardiopulmonary bypass. Acute kidney injury is defined according to the KIDIGO guidelines.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
serum and urine metabolome studies | January 2025 - December 2025
  The preoperative and postoperative metabolomic differences in blood and urine between AKI group and non-AKI group were compared.

CONTACTS AND LOCATIONS:
Overall Officials: Chen Wenxiu, Principal Investigator — Nanjing First Hospital, Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing, China